CLINICAL TRIAL: NCT01835756
Title: A Double-Blind, Placebo-Controlled Randomized Evaluation of the Effect of the Erchonia ML Scanner (MLS) on Low Back Pain Clinical Study
Brief Title: Study of Low Level Laser Therapy to Treat Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_LBP_01
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erchonia MLS (Active Comparator): The Erchonia® MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light.
  Interventions: Device: Erchonia MLS
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia MLS but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia MLS — The Erchonia® MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light. The Erchonia MLS is applied to the lower back and hips area for 15 minutes per treatment administration, 6 times across 3 weeks, 2 times per week.
  Arms: Erchonia MLS
Device: Placebo Laser — The Placebo Laser has the same appearance and administration application as the Erchonia MLS but does not emit any therapeutic light.
  Arms: Placebo Laser

SUMMARY:
The purpose of this study is to determine whether the Erchonia® ML Scanner (MLS) is effective in the treatment of acute minor episodic chronic low back pain of musculoskeletal origin.

DETAILED DESCRIPTION:
Back pain is a common musculoskeletal disorder affecting 80% of people at some point in their lives. It is the second most common neurological ailment in the United States, second only to headache, and it is the most common cause of job-related disability and a leading contributor to missed work. Around $50 billion is spent in the U.S. each year to treat low back pain. Men and women are equally affected, with the most common age affected being between 30 and 50 years.

Most low back pain stems from benign musculoskeletal problems, referred to as non-specific low back pain, which is the etiology being evaluated in this study. It is caused by lumbar sprain or strain a stretch injury to the ligaments, tendons, and/or muscles of the low back.

Current mainstream treatment approaches for low back pain due to lumbar sprain strain focus on reducing pain and inflammation, including rest; oral and topical over-the-counter and prescription medications; local heat applications; massage and exercise. Alternative treatment options include acupuncture; chiropractic manipulation; biofeedback; traction; transcutaneous electrical nerve stimulation (TENS); and ultrasound. Surgical procedures are also a treatment option for low back pain, and although the outcomes are often poor and do not last, back surgery remains the 3rd most common form of surgery in the United States, with about 300,000 back surgeries performed annually.

Low Level Laser Therapy (LLLT) communicates information to the receptors on the membrane of the cell and mitochondrion (the enzymatic engine of the cell). This energetic information reaches the cell's DNA, which directly controls cell function. When the cells receive better information, they work better, as do the tissues they comprise, like bones, cartilage, tendons, ligaments, etc. In this way, LLLT promotes the healing and regeneration of damaged tissues, having both local effects on tissue function and also systemic effects carried throughout the body by the blood and acupuncture meridians. The key basic physiological effects of low level laser light include increased cell membrane polarization and permeability; Adenosine-5-triphosphate (ATP) production and respiratory chain activity; enzyme activity; collagen and epithelial production; capillary formation; macrophage (immune) activity; analgesic effects due to elevated endorphin production, electrolytic nerve blockage, and improved blood and lymph flow; anti-inflammatory effect due to improved circulation and accelerated tissue regeneration; and increased production of antioxidants. Of additional benefit is that light energy from low level lasers will only be absorbed by cells and tissues that are not functioning normally and has no effect on healthy cells.

Therefore, low level laser therapy has the potential benefit of providing an effective means of reducing low back pain that is simple, quick, non-invasive and side-effect free.

ELIGIBILITY:
Inclusion Criteria:

* Primary pain is in the lower back
* Low back pain is of musculoskeletal origin stemming from benign musculoskeletal problems wherein the etiology is lumbar sprain or strain
* Diagnosis based on review of patient history, physical examination, medication use history and review of prior medical records
* Low back pain is episodic chronic, having occurred and recurred over regular or irregular intervals of time over at least the last 3 months
* Degree of Pain rating on the visual analog scale (VAS) is 40 or greater
* Subject is willing and able to refrain from taking non study medications and herbal supplements for the relief of pain or inflammation including muscle relaxants throughout study participation
* Subject is willing and able to refrain from non study procedure therapies for the management of low back pain throughout study participation
* Primary language is English

Exclusion Criteria:

* Low back pain is undiagnosed or has been diagnosed as being other than of benign musculoskeletal origin wherein the etiology is lumbar sprain or strain
* Low back pain has been diagnosed or cannot be satisfactorily ruled out as being in whole or in part due to one or more of the following origins - mechanical, inflammatory, neoplastic, metabolic origin, psychosomatic
* Tension myositis syndrome
* Known herniated disc injury
* Osteoporosis with compression fractures
* Congenital deformity of spine
* Current active chronic pain disease
* Cancer or cancer treatment in the past 6 months
* Use of the following analgesics within 7 days of study onset - paracetamol, acetominophen, non-steroidal anti-inflammatory drugs (NSAIDs), compound analgesics, topical analgesics
* Use of the following muscle relaxants within the prior 30 days of study onset - cyclobenzaprine, diazepam, meprobamate
* Use of the following muscle relaxants within 7 days of study onset - carisoprodol, Metaxalone
* Use of the following antidepressants within 30 days of study onset if consumption has commenced within that 30 day period - duloxetine, amitriptyline, imipramine, clomipramine, nortriptyline, desipramine, selective serotonin reuptake inhibitors (SSRIs)
* Systemic corticosteroid therapy or narcotics taken within 30 days (inhaled and topical corticosteroids okay) of study onset
* Local or epidural injection of corticosteroids within 3 months of study onset
* Botulinum toxin injection for chronic low back pain within 4 months of study onset
* Active infection, wound, other external trauma to the treatment area
* Surgery to the lower back or spine in the past 12 months
* Medical, physical or other contraindications for, or sensitivity to, light therapy
* Pregnant, breast feeding or planning pregnancy prior to study end
* Serious mental health illness such as dementia or schizophrenia or psychiatric hospitalization in past 2 years
* Developmental disability or cognitive impairment that precludes adequate comprehension of consent form or the ability to record study measurements
* Participation in other research in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor Berry, DC, Principal Investigator; Mark B Burdorf, DC, DACNB, Principal Investigator
Locations (2):
- United States (2):
  - South Mountain Chiropractic Center, Chandler, Arizona
  - Mark B. Burdorf DC, Scottsdale, Arizona

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia MLS: The Erchonia MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light. It is applied to the lower back and hips area for 30 minutes per treatment administration, 6 times across 3 weeks, 2 times per week.
Period: Overall Study
Arm/Group | Erchonia MLS | Placebo Laser
Started | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erchonia MLS: The Erchonia MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light. The Erchonia MLS is applied to the lower back and hips area for 15 minutes per treatment administration, 6 times across 3 weeks, 2 times per week.
- Placebo Laser: The Placebo Laser has the same appearance and treatment application as the Erchonia MLS but does not emit any therapeutic light.
- Total: Total of all reporting groups
Arm/Group | Erchonia MLS | Placebo Laser | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.90 (12.62) | 49.48 (16.39) | 51.69 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 29
  Male | 15 | 18 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 30 | 27 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62
Duration of Low Back Pain [Mean (Standard Deviation); unit: months] — Duration of low back pain was recorded as the number of months the subject reporting experiencing ongoing low back pain.
  months | 92.65 (95.42) | 93.45 (110.86) | 93.05 (102.60)
Visual Analog Scale (VAS) Degree of Low Back Pain Rating [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Pain Scale (VAS) is one of the three most commonly used scales for assessing chronic pain. The VAS scale ranges from 0 to 100 mm, with 0 indicating no pain and 100 indicating the worst pain imaginable. The subject marks on the line the spot for the pain intensity, which is then measured using a ruler.
  units on a scale | 61.19 (13.24) | 55.94 (10.74) | 58.56 (12.35)

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Proportion of Primary Outcome Successes Between Treatment Groups
Description: Primary outcome success for an individual subject was defined as a 30% or greater change (decrease) in VAS pain score at 4 months post-procedure relative to baseline. The VAS is a straight line scale that is marked on one end with a '0' for 'no pain' and at the other end with '100' for 'worse pain imaginable.' A higher score indicates a greater level of pain, and a lower score indicates a lower level of pain. A negative (-) percent change in VAS rating indicates a decrease in pain level and is positive for individual subject success. A positive (+) percent change indicates an increase in pain level and is negative for individual subject success. Overall study success was defined as a 35% or greater difference in the proportion of individual primary outcome successes in each treatment group, in favor of the active treatment group.
Time Frame: 4 Months
Measure: Number; unit: participants
Groups:
- Erchonia MLS: The Erchonia MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light, applied to the lower back and hips area for 15 minutes per treatment administration, 6 times across 3 weeks, 2 times per week.
- Placebo Laser: The Placebo Laser has the same appearance and administration application as the active Erchonia MLS but does not emit any therapeutic light.
Arm/Group | Erchonia MLS | Placebo Laser
Number analyzed (Participants) | 31 | 31
participants | 27 | 9
Statistical Analysis 1: Comparison: Erchonia MLS vs Placebo Laser; Test type: Superiority or Other; p < 0.00001, t-test, 2 sided

2. Secondary Outcome: Change in Low Back Pain Visual Analog Scale (VAS) Score
Description: The VAS is a straight line scale that is marked on one end with a '0' for 'no pain' and at the other end with '100' for 'worse pain imaginable.' A higher score on the VAS indicates a greater level of pain, and a lower score indicates a lower level of pain.A decrease in the VAS pain rating indicates a reduction in low back pain and is positive for study success. An increase in the VAS pain rating indicates a worsening of low back pain and is negative for study success. The mean change in low back pain score recorded on the Visual Analog Scale (VAS) from baseline to 4 months post-procedure was calculated for each treatment group.
Time Frame: Baseline and 4 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia MLS | Placebo Laser
Number analyzed (Participants) | 31 | 31
units on a scale | -39.32 (22.50) | -5.52 (20.17)
Statistical Analysis 1: Comparison: Erchonia MLS vs Placebo Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Satisfaction With Study Outcome
Description: At study endpoint, the subject was asked to rate how satisfied he or she was with any overall change in low back pain attained following the procedure administration phase with the Erchonia MLS Laser, using the following five-point scale:
  Very Satisfied Somewhat Satisfied Neither Satisfied nor Dissatisfied Not Very Satisfied Not at All Satisfied
  Results are reported as the number of subjects who reported being 'Very Satisfied' or 'Somewhat Satisfied' with the study outcome.
Time Frame: 4 Months
Measure: Number; unit: participants
Arm/Group | Erchonia MLS | Placebo Laser
Number analyzed (Participants) | 31 | 31
participants | 26 | 7

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Erchonia MLS: The Erchonia MLS contains 10 independent diodes, each emitting 17 milliwatts (mW), 635 nanometers (nm) of red laser light applied to the lower back and hips area for 30 minutes per treatment administration, 6 times across 3 weeks, 2 times per week.
Arm/Group | Erchonia MLS | Placebo Laser
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No